CLINICAL TRIAL: NCT02148952
Title: A Matched-pair, Cluster Randomized Trial to Measure the Efficacy of the WHO Safe Childbirth Checklist Program on Severe Maternal, Fetal and Newborn Harm
Brief Title: BetterBirth: A Trial of the WHO Safe Childbirth Checklist Program
Acronym: BetterBirth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: World Health Organization (Other); Population Services International (Other); Jawaharlal Nehru Medical College (Other); Community Empowerment Lab (Other); Brigham and Women's Hospital (Other); Bill and Melinda Gates Foundation (Other); MacArthur Foundation (Other)
Responsible Party: Principal Investigator, Katherine Semrau, Principal Investigator, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HSPH OPP1017378
Record Dates: First submitted 2014-02-13; First posted 2014-05-29 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Maternal Death; Maternal Morbidity; Stillbirth; Neonatal Death
Keywords: Maternal Health; Maternal Death; Maternal Morbidity; Stillbirth; Neonatal Mortality; Quality Improvement; Resource Limited Settings; Checklist; Safe Childbirth
MeSH Terms: conditions — Maternal Death; Stillbirth; Perinatal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Health Facility (Experimental): WHO Safe Childbirth Checklist Program
  Interventions: Behavioral: WHO Safe Childbirth Checklist Program
- Control Health Facility (No Intervention): Matched control facilities providing comparison for intervention facilities

INTERVENTIONS:
Behavioral: WHO Safe Childbirth Checklist Program — The IHF group will receive the WHO Safe Childbirth Checklist Program designed to maximize likelihood of effective and sustained uptake of the program by birth attendants in the designated facilities. The program includes three key implementation steps that involve: engagement of leadership and clinicians at the state, district, and local levels, a formal launch to introduce the Checklist, and support through peer coaching and data feedback. The intervention facilities will also receive a standardized maternity register to ensure appropriate data collection.
  Arms: Intervention Health Facility

SUMMARY:
The purpose of this study is to measure the impact of a checklist-based childbirth safety program (the WHO Safe Childbirth Checklist Program) on reduction of severe maternal, fetal, and newborn harm in institutional deliveries in north India.

DETAILED DESCRIPTION:
The WHO Safe Childbirth Checklist Program is a quality improvement program designed to support health workers to deliver evidence-based practices to women and newborns around the time of institutional childbirths. At the program's core is the Safe Childbirth Checklist, a 31-item list of essential practices that target the major causes of maternal and newborn mortality in low-resource settings globally. The program was developed over 3 years by a partnership of WHO and HSPH, working with a large international network of experts and stakeholders in maternal, fetal, and newborn health. Pilot testing of the program at a public-sector birth center in south India demonstrated dramatic improvements in health worker adherence to essential childbirth-related clinical care standards. The current study is a matched-pair, cluster randomized trial to measure the efficacy of the program in reducing severe maternal and newborn harm. This trial will be conducted at approximately 120 health facilities in Uttar Pradesh, India.

ELIGIBILITY:
Inclusion Criteria:

* For measuring outcomes, inclusion criteria are all mothers admitted to a study site for childbirth and newborn babies who are to be followed-up. In case a mother or baby from an enrolled site is referred out to another facility (before or after delivery) the mother-baby dyad will be included in the study and the outcome will be allocated to the referring facility
* For a smaller subset of birth events (approximately 4,650 deliveries total), health worker practices will be observed to measure the impact of the SCC program on delivery of essential practices, as a secondary outcome. A convenience sample of women who agree to observation and their babies cared for by the health workers around the time of childbirth at the facility during data collectors' duty hours will be included in this component of the study.

Exclusion Criteria:

* Mothers who have been referred into the facility by an inter-facility transfer.
* Mothers being managed for abortion.
* Mothers who refuse consent for follow-up

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 157689 (Actual)
Dates: Start 2014-11; Primary Completion 2017-01-20 (Actual); Study Completion 2017-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atul Gawande, MD, MPH, Principal Investigator — Harvard School of Public Health (HSPH); Vishwajeet Kumar, MBBS, MPH, Principal Investigator — Community Empowerment Lab; Bhala Kodkany, MBBS, Principal Investigator — Jawarhlal Nehru Medical College; Katherine Semrau, PhD, Principal Investigator — Harvard Medical School/ Ariadne Labs
Locations (1):
- PSI, Lucknow, Uttar Pradesh, India

REFERENCES:
- [Derived] Lofgren KT, Bobanski L, Tuller DE, Singh VP, Marx Delaney M, Jurczak A, Ragavan M, Kalita T, Karlage A, Resch SC, Semrau KEA. Estimating maternity ward birth attendant time use in India: a microcosting study. BMJ Open. 2022 Feb 7;12(2):e054164. doi: 10.1136/bmjopen-2021-054164. PMID 35131826
- [Derived] Semrau KE, Miller KA, Lipsitz S, Fisher-Bowman J, Karlage A, Neville BA, Krasne M, Gass J, Jurczak A, Pratap Singh V, Singh S, Marx Delaney M, Hirschhorn LR, Kodkany B, Kumar V, Gawande AA. Does adherence to evidence-based practices during childbirth prevent perinatal mortality? A post-hoc analysis of 3,274 births in Uttar Pradesh, India. BMJ Glob Health. 2020 Sep;5(9):e002268. doi: 10.1136/bmjgh-2019-002268. PMID 32928798
- [Derived] Barnhart DA, Semrau KEA, Zigler CM, Molina RL, Delaney MM, Hirschhorn LR, Spiegelman D. Optimizing the development and evaluation of complex interventions: lessons learned from the BetterBirth Program and associated trial. Implement Sci Commun. 2020 Feb 25;1:29. doi: 10.1186/s43058-020-00014-8. eCollection 2020. PMID 32885188
- [Derived] Molina RL, Neal BJ, Bobanski L, Singh VP, Neville BA, Delaney MM, Lipsitz S, Karlage A, Shetye M, Semrau KEA. Nurses' and auxiliary nurse midwives' adherence to essential birth practices with peer coaching in Uttar Pradesh, India: a secondary analysis of the BetterBirth trial. Implement Sci. 2020 Jan 3;15(1):1. doi: 10.1186/s13012-019-0962-7. PMID 31900167
- [Derived] Hirschhorn LR, Krasne M, Maisonneuve J, Kara N, Kalita T, Henrich N, Rana D, Maji P, Delaney MM, Firestone R, Sharma N, Kumar V, Gawande AA, Semrau KEA. Integration of the Opportunity-Ability-Motivation behavior change framework into a coaching-based WHO Safe Childbirth Checklist program in India. Int J Gynaecol Obstet. 2018 Sep;142(3):321-328. doi: 10.1002/ijgo.12542. Epub 2018 Jun 20. PMID 29862506
- [Derived] Maisonneuve JJ, Semrau KEA, Maji P, Pratap Singh V, Miller KA, Solsky I, Dixit N, Sharma J, Lagoo J, Panariello N, Neal BJ, Kalita T, Kara N, Kumar V, Hirschhorn LR. Effectiveness of a WHO Safe Childbirth Checklist Coaching-based intervention on the availability of Essential Birth Supplies in Uttar Pradesh, India. Int J Qual Health Care. 2018 Dec 1;30(10):769-777. doi: 10.1093/intqhc/mzy086. PMID 29718354
- [Derived] Semrau KEA, Hirschhorn LR, Marx Delaney M, Singh VP, Saurastri R, Sharma N, Tuller DE, Firestone R, Lipsitz S, Dhingra-Kumar N, Kodkany BS, Kumar V, Gawande AA; BetterBirth Trial Group. Outcomes of a Coaching-Based WHO Safe Childbirth Checklist Program in India. N Engl J Med. 2017 Dec 14;377(24):2313-2324. doi: 10.1056/NEJMoa1701075. PMID 29236628
- [Derived] Gass JD Jr, Misra A, Yadav MNS, Sana F, Singh C, Mankar A, Neal BJ, Fisher-Bowman J, Maisonneuve J, Delaney MM, Kumar K, Singh VP, Sharma N, Gawande A, Semrau K, Hirschhorn LR. Implementation and results of an integrated data quality assurance protocol in a randomized controlled trial in Uttar Pradesh, India. Trials. 2017 Sep 7;18(1):418. doi: 10.1186/s13063-017-2159-1. PMID 28882167
- [Derived] Semrau KE, Hirschhorn LR, Kodkany B, Spector JM, Tuller DE, King G, Lipsitz S, Sharma N, Singh VP, Kumar B, Dhingra-Kumar N, Firestone R, Kumar V, Gawande AA. Effectiveness of the WHO Safe Childbirth Checklist program in reducing severe maternal, fetal, and newborn harm in Uttar Pradesh, India: study protocol for a matched-pair, cluster-randomized controlled trial. Trials. 2016 Dec 7;17(1):576. doi: 10.1186/s13063-016-1673-x. PMID 27923401
- See also: WHO Safe Childbirth Checklist — https://www.who.int/teams/integrated-health-services/patient-safety/research/safe-childbirth
- See also: Ariadne Labs — http://www.ariadnelabs.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 320 facilities were assessed for eligibility. 200 were excluded (37 did not meet inclusion criteria, 163 did not have a matching facility identified).
  A total of 163,939 women were screened for eligibility; of those, 161,107 women were eligible for participation, and 157,689 women consented and were enrolled into the trial.
Units Other Than Participants: facilities
Groups:
- Intervention Health Facility Participants: Women at intervention facilities who registered for labor and delivery, eligible for inclusion, and who provided consent.
  Intervention Health Facilities received the WHO Safe Childbirth Checklist Program.
  WHO Safe Childbirth Checklist Program: The IHF group will receive the WHO Safe Childbirth Checklist Program designed to maximize likelihood of effective and sustained uptake of the program by birth attendants in the designated facilities. The program includes three key implementation steps that involve: engagement of leadership and clinicians at the state, district, and local levels, a formal launch to introduce the Checklist, and support through peer coaching and data feedback. The intervention facilities will also receive a standardized maternity register to ensure appropriate data collection.
- Control Health Facility Participants: Women at control health facilities who registered for labor and delivery, eligible for inclusion, and who provided consent.
  Matched control facilities provided comparison for intervention facilities.
Period: Assessing Eligibility and Consent
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Started (This includes all women who registered for delivery.) | 83166; 60 facilities | 80773; 60 facilities
Completed (This includes all women who were eligible for inclusion and consented to follow-up.) | 80063; 60 facilities | 77626; 60 facilities
Not Completed | 3103; 0 facilities | 3147; 0 facilities
Not completed — Were not eligible for inclusion | 1241 | 1591
Not completed — Did not consent or declined follow-up | 1862 | 1556
Period: Follow-Up
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Started | 80063; 60 facilities | 77626; 60 facilities
Completed | 79798; 60 facilities | 77347; 60 facilities
Not Completed | 265; 0 facilities | 279; 0 facilities
Not completed — Lost to Follow-up | 219 | 231
Not completed — Withdrawal by Subject | 46 | 48

BASELINE CHARACTERISTICS:
Population: The baseline analysis population may refer to number of women, number of newborns, or number of facilities, depending on the measure. We obtained facility consent to collect baseline information for a total of 161,107 women who were eligible for inclusion. A total of 157,687 women consented to participate in follow-up.
Units Other Than Participants: Facilities
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants | Total
Number analyzed (Participants) | 81,925 | 79,182 | 161107
Number analyzed (Facilities) | 60 | 60 | 120
Age, Continuous [Mean (Full Range); unit: years] — Please note the measure of dispersion is a 95% confidence interval (not full range).
  years | 25.6 [25.5 to 25.8] | 25.7 [25.5 to 25.9] | 25.66 [25.54 to 25.79]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex of the newborn. Population: This refers to the number of newborns whose mothers were enrolled in the trial. In "unknown" cases, the mother was referred to another facility before the data were captured.
  Participants
    number analyzed (Participants) | 81447 | 78663 | 160110
    Sex of newborn: Male | 40558 | 39063 | 79621
    Sex of newborn: Female | 36976 | 36266 | 73242
    Sex of newborn: Unknown | 3913 | 3334 | 7247
Sex: Female, Male [Count of Participants; unit: Participants] — Pregnant women were enrolled in the trial; thus, all are female.
  Participants
    Female | 81925 | 79182 | 161107
    Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: participants]
  India | 81925 | 79182 | 161107
Mean Annual Delivery Load [Mean (Full Range); unit: deliveries] — This characteristic was used for facility matching before randomization. Please note the measure of dispersion is a 95% confidence interval (not full range).
  deliveries | 1599 [1486 to 1712] | 1683 [1552 to 1814] | 1641 [1531 to 1751]
Functional Classification [Count of Units; unit: Facilities] — This characteristic was used for facility matching before randomization.
  Facilities
    Primary health center | 23 | 23 | 46
    Community Health Center | 27 | 29 | 56
    First referral unit | 10 | 8 | 18
Mean distance to district hospital [Mean (Full Range); unit: km] — This characteristic was used for facility matching before randomization. Please note the measure of dispersion is a 95% confidence interval (not full range).
  km | 29.5 [25.9 to 33.1] | 30.3 [27.2 to 33.4] | 29.9 [27.0 to 32.8]
Mean skilled birth attendants per facility [Mean (Full Range); unit: number of skilled birth attendants] — This characteristic was used for facility matching before randomization. Please note the measure of dispersion is a 95% confidence interval (not full range).
  number of skilled birth attendants | 4.4 [4.1 to 4.7] | 4.4 [4.1 to 4.7] | 4.4 [4.1 to 4.7]
Cluster Size [Mean (Full Range); unit: participants per site] — Cluster size is the total number of pregnant women enrolled per site (cluster). Please note the measure of dispersion is a 95% confidence interval (not full range).
  participants per site | 1365 [515 to 2697] | 1320 [646 to 2198] | 1343 [1261 to 1423]
Mean previous pregnancies [Mean (Full Range); unit: previous pregnancies] — Please note the measure of dispersion is a 95% confidence interval (not full range).
  previous pregnancies | 2.4 [2.3 to 2.4] | 2.3 [2.3 to 2.4] | 2.36 [2.32 to 2.39]
Minutes between admission and delivery [Mean (Full Range); unit: minutes] — Please note the measure of dispersion is a 95% confidence interval (not full range).
  minutes | 200 [184 to 216] | 206 [191 to 220] | 203 [192 to 213]
Providers attending delivery [Count of Participants; unit: Participants]
  Doctor: number analyzed (Participants) | 81925 | 79,182 | 161107
  Doctor | 11115 | 11599 | 22714
  Nurse | 66687 | 64117 | 130804
  Auxiliary nurse midwife | 15311 | 14549 | 29860
  Others | 2633 | 6560 | 9193
No. of offspring [Count of Participants; unit: Participants]
  Singleton | 80402 | 77582 | 157984
  Sets of twins | 515 | 533 | 1048
  Sets of triplets | 5 | 5 | 10
  Unknown | 1,003 | 1,062 | 2065
Low birth weight [Count of Participants; unit: Participants] — Occurrence of low birth weight. Low birth weight was defined as 2500 g or less. Population: This refers to the number of newborns whose mothers were enrolled in the trial.
  Participants
    number analyzed (Participants) | 81447 | 78663 | 160110
    (all) | 22316 | 22728 | 45044
Preterm birth [Count of Participants; unit: Participants] — Occurrence of preterm birth. Preterm birth was defined as fewer than 37 weeks of gestation. Population: This refers to the number of newborns whose mothers were enrolled in the trial.
  Participants
    number analyzed (Participants) | 81447 | 78663 | 160110
    (all) | 15941 | 17703 | 33644

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Composite Measure of Perinatal Death, Maternal Death, or Maternal Severe Complications Within 7 Days
Description: The primary outcome was a composite outcome of events occurring within the first 7 days after delivery, incorporating stillbirth; early neonatal death; maternal death; or self-reported maternal severe complications, including seizures, loss of consciousness for more than 1 hour, fever with foul-smelling vaginal discharge, hemorrhage, or stroke.
Time Frame: 0-7 days after delivery
Population: The denominator for this analysis is all women who had non-missing information about their death, their baby(s) and their morbidity.
Measure: Number; unit: percentage of women/newborn dyads
Groups:
- Intervention Health Facility Participants: Women/newborn dyads at intervention facilities who registered for labor and delivery, eligible for inclusion, and who provided consent.
  Intervention Health Facilities received the WHO Safe Childbirth Checklist Program.
  WHO Safe Childbirth Checklist Program: The IHF group will receive the WHO Safe Childbirth Checklist Program designed to maximize likelihood of effective and sustained uptake of the program by birth attendants in the designated facilities. The program includes three key implementation steps that involve: engagement of leadership and clinicians at the state, district, and local levels, a formal launch to introduce the Checklist, and support through peer coaching and data feedback. The intervention facilities will also receive a standardized maternity register to ensure appropriate data collection.
- Control Health Facility Participants: Women/newborn dyads at control health facilities who registered for labor and delivery, eligible for inclusion, and who provided consent.
  Matched control facilities provided comparison for intervention facilities.
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 79334 | 76897
percentage of women/newborn dyads | 15.1 | 15.3
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Test type: Superiority — We hypothesized a 15% reduction in the composite outcome between the intervention and control arm; p = 0.90, Chi-squared, Corrected; In secondary analyses, a Rao-Scott test with 3 degrees of freedom resulted in a p value of 0.88; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.83 to 1.18] — Relative risks are for the intervention group as compared with the control group and are adjusted for clustering and matching. The denominators shift owing to missing data on outcomes

2. Secondary Outcome: Percentage of Participants With Perinatal Death or Maternal Death Within 7 Days
Description: Percentage of participants with composite rate of perinatal death and maternal death within 7 days
Time Frame: 0-7 days after delivery
Population: The denominator for this analysis is all women who had non-missing information about their death, and their baby(s)
Measure: Number; unit: percentage of women and newborns
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 79789 | 77337
percentage of women and newborns | 4.9 | 4.7
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Test type: Superiority; p = 0.67, Chi-squared, Corrected; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.89 to 1.20] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Count of Participants With Perinatal Death Within 7 Days
Description: Count of participants with perinatal death within 7 days (combined stillbirth or neonatal death)
Time Frame: 0-7 days
Population: There is a discrepancy between the denominator of each primary and secondary outcome because there were a different number of newborns than mothers in the trial. Additionally, we do not have data on every participant for every question. As such, the denominator is specific for each outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 79790 | 77338
Participants | 3839 | 3606
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Test type: Superiority; p = 0.68, Chi-squared, Corrected; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.89 to 1.20]

4. Secondary Outcome: Count of Participants With Stillbirth
Description: Newborn outcome; rate of stillbirth
Time Frame: 0-7 days after delivery
Population: The denominator for this analysis is all women who had non-missing information about whether their baby(s) experienced stillbirth.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 80061 | 77454
Participants | 1513 | 1559
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Test type: Superiority; p = 0.56, Chi-squared, Corrected; Risk Ratio (RR) = 0.94, 95% CI 2-sided [0.76 to 1.16] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Count of Participants With Early Neonatal Death
Description: Newborn outcome; rate of early neonatal death
Time Frame: 0-7 days after delivery
Population: The denominator for this analysis is all women who had non-missing information about whether their baby(s) experienced neonatal death.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 78360 | 75851
Participants | 2409 | 2119
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Test type: Superiority; p = 0.19, Chi-squared, Corrected; Risk Ratio (RR) = 1.10, 95% CI 2-sided [0.95 to 1.27]

6. Secondary Outcome: Count of Participants With Maternal Death
Description: Maternal outcome; rate of maternal death
Time Frame: 0-7 days after delivery
Population: The denominator for this analysis is all women who had non-missing information about maternal death status.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 79,797 | 77,346
Participants | 78 | 71
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Test type: Superiority; p = 0.73, Chi-squared, Corrected; Risk Ratio (RR) = 1.11, 95% CI 2-sided [0.74 to 1.53] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Count of Participants With Severe Maternal Complications
Description: Maternal outcome; any severe maternal complication within 7 days
Time Frame: 0-7 days after delivery
Population: The denominator for this analysis is all women who had non-missing information about each morbidity. Not every respondent answered each question, so each row has a different denominator. Only women who answered all specific morbidity questions were incorporated into the participant count for "any maternal severe complication within 7 days".
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 79706 | 77257
Participants
  Any maternal severe complication within 7 days: number analyzed (Participants) | 79342 | 76907
  Any maternal severe complication within 7 days | 9086 | 9037
  Seizures | 67 | 70
  Loss of consciousness for >1 hour: number analyzed (Participants) | 79649 | 77196
  Loss of consciousness for >1 hour | 505 | 493
  High fever with foul-smelling vaginal discharge: number analyzed (Participants) | 79459 | 77018
  High fever with foul-smelling vaginal discharge | 4073 | 3871
  Hemorrhage: number analyzed (Participants) | 79648 | 77198
  Hemorrhage | 5745 | 5875
  Stroke: number analyzed (Participants) | 79703 | 77257
  Stroke | 9 | 12
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Rate any severe maternal complication within 7 days; Test type: Superiority; p = 0.81, Chi-squared, Corrected; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.79 to 1.20] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Rate of seizures; Test type: Superiority; p = 0.76, Chi-squared, Corrected; Risk Ratio (RR) = 0.89, 95% CI 2-sided [0.57 to 1.52] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Rate of loss of consciousness for > 1 hr; Test type: Superiority; p = 0.97, Chi-squared, Corrected; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.70 to 1.41] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Rate of high fever with foul-smelling vaginal discharge; Test type: Superiority; p = 0.90, Chi-squared, Corrected; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.76 to 1.38] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Rate of hemorrhage; Test type: Superiority; p = 0.61, Chi-squared, Corrected; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.77 to 1.17] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Rate of stroke; Test type: Superiority; p = 0.41, Chi-squared, Corrected; Risk Ratio (RR) = 0.50, 95% CI 2-sided [0.34 to 1.58] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Count of Participants With Cesarean Section
Description: Rate of cesarean section
Time Frame: Around the time of delivery during facility stay, an expected average of 2 days (although individual patients may vary)
Population: The denominator for this analysis is all women who had non-missing information about whether they had a cesarean section.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 80922 | 78120
Participants | 1469 | 1330
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Test type: Superiority; p = 0.74, Chi-squared, Corrected; Risk Ratio (RR) = 1.07, 95% CI 2-sided [0.72 to 1.58]

9. Secondary Outcome: Count of Participants With Maternal Referral, Before or After Delivery
Description: Maternal outcome; Rate of maternal inter-facility transfer
Time Frame: 0-7 days after delivery
Population: The denominator for this analysis is all women who had non-missing information about their status regarding referral before and after delivery.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 81925 | 79182
Participants | 5381 | 4779
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Test type: Superiority; p = 0.57, Chi-squared, Corrected; Risk Ratio (RR) = 1.09, 95% CI 2-sided [0.81 to 1.47] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Count of Participants With Newborn Referral
Description: Newborn outcome; Newborn referral
Time Frame: 0-7 days after delivery
Population: The denominator for this analysis is all women who had non-missing information about their newborn(s) referral status.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 81925 | 79182
Participants | 1455 | 1186
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Test type: Superiority; p = 0.41, Chi-squared, Corrected; Risk Ratio (RR) = 1.19, 95% CI 2-sided [0.78 to 1.80] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Count of Participants With Hysterectomy Within 7 Days
Description: Rate of hysterectomy within 7 days
Time Frame: 0-7 days after delivery
Population: The denominator for this analysis is all women who had non-missing information about their hysterectomy status within 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 79705 | 77252
Participants | 19 | 18
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Test type: Superiority; p = 0.95, Chi-squared, Corrected; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.45 to 2.13] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Count of Participants With Blood Transfusion Within 7 Days
Description: Rate of blood transfusion within 7 days
Time Frame: 0-7 days after delivery
Population: The denominator for this analysis is all women who had non-missing information about their status regarding blood transfusion within 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 79697 | 77254
Participants | 640 | 625
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Test type: Superiority; p = 0.97, Chi-squared, Corrected; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.69 to 1.43]

13. Secondary Outcome: Count of Mothers Returning to Facility for a Health Problem Within 7 Days
Description: Maternal Outcome; Rate of need for follow-up care for Mother
Time Frame: 0-7 days after delivery
Population: The denominator for this analysis is all women who had non-missing information about returning to a health facility for a health problem within 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 79655 | 77220
Participants | 2014 | 2141
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Test type: Superiority; p = 0.32, Chi-squared, Corrected; Risk Ratio (RR) = 0.91, 95% CI 2-sided [0.76 to 1.10] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Count of Newborns Returning to Facility for a Health Problem Within 7 Days
Description: Newborn outcome; Rate of need for follow-up care for newborn (or at least one newborn in case of twins)
Time Frame: 0-7 days after delivery
Population: The denominator for this analysis is all women who had non-missing information about status of at least one baby returning to the facility for a health problem within 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 77419 | 75117
Participants | 4474 | 4722
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Test type: Superiority; p = 0.30, Chi-squared, Corrected; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.78 to 1.08] — [estimate comment as in outcome 1, analysis 1]

15. Other Pre Specified Outcome: Mean Number of 18 Essential Birth Practices Performed at 2 Months Post-intervention Start
Description: Birth attendant's rate of completion of "Process measures" resulting from Safe Childbirth Checklist program will be assessed in a sample of total birth events at 2 months after the intervention is introduced to intervention facilities. The below measures reflect the mean number of 18 essential birth practices performed across the intervention versus control facilities at 2 months post-intervention start.
Time Frame: 2 months post-intervention start
Population: The denominator for this analysis is all women who were observed for at least one pause point 2 months post-intervention start in the site.
Measure: Mean (95% Confidence Interval); unit: essential birth practices performed
Groups:
- Intervention Health Facility Participants: Women/newborn dyads at intervention facilities who registered for labor and delivery, eligible for inclusion, and who provided consent for observation.
  Intervention Health Facilities received the WHO Safe Childbirth Checklist Program.
  WHO Safe Childbirth Checklist Program: The IHF group will receive the WHO Safe Childbirth Checklist Program designed to maximize likelihood of effective and sustained uptake of the program by birth attendants in the designated facilities. The program includes three key implementation steps that involve: engagement of leadership and clinicians at the state, district, and local levels, a formal launch to introduce the Checklist, and support through peer coaching and data feedback. The intervention facilities will also receive a standardized maternity register to ensure appropriate data collection.
- Control Health Facility Participants: Women/newborn dyads at control health facilities who registered for labor and delivery, eligible for inclusion, and who provided consent for observation.
  Matched control facilities provided comparison for intervention facilities.
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 1259 | 1304
essential birth practices performed | 13.1 [12.1 to 14.0] | 7.5 [6.9 to 8.1]
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Other = 0

16. Other Pre Specified Outcome: Count of Participants Where Essential Birth Practices Were Observed at Admission, 2 Months Post-intervention Start
Description: Birth attendant's rate of completion of "Process measures" resulting from Safe Childbirth Checklist program will be assessed in a sample of total birth events at 2 months after the intervention is introduced to intervention facilities. The below measures reflect the essential birth practices performed at the time of the woman's admission to the facility, 2 months post-intervention start.
Time Frame: 2 months post-intervention start
Population: The denominator for this analysis is all women who were observed at admission, 2 months post-intervention start in the site.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Health Facility Participants: Women at intervention facilities who registered for labor and delivery, were eligible for inclusion, and who provided consent for observation.
  Intervention Health Facilities received the WHO Safe Childbirth Checklist Program.
  WHO Safe Childbirth Checklist Program: The IHF group will receive the WHO Safe Childbirth Checklist Program designed to maximize likelihood of effective and sustained uptake of the program by birth attendants in the designated facilities. The program includes three key implementation steps that involve: engagement of leadership and clinicians at the state, district, and local levels, a formal launch to introduce the Checklist, and support through peer coaching and data feedback. The intervention facilities will also receive a standardized maternity register to ensure appropriate data collection.
- Control Health Facility Participants: Women at control facilities who registered for labor and delivery, were eligible for inclusion, and who provided consent for observation.
  Matched control facilities provided comparison for intervention facilities.
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 1048 | 1090
Participants
  Birth companion present | 1048 | 1087
  Maternal blood pressure taken | 606 | 64
  Maternal temperature taken | 569 | 4
  Partography started | 10 | 1
  Checklist use | 595 | 1
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Birth Companion Present; Test type: Superiority; p = 0.18, Chi-squared, Corrected; Other = 0 — The relative risk could not be calculated owing to 100% or 0% values in one group
Statistical Analysis 2: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Maternal blood pressure taken; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 9.8, 95% CI 2-sided [3.4 to 28.3]
Statistical Analysis 3: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Maternal temperature taken; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 132, 95% CI 2-sided [26.9 to 645]
Statistical Analysis 4: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Partography started; Test type: Superiority; p = 0.01, Chi-squared, Corrected; Risk Ratio (RR) = 7.3, 95% CI 2-sided [1.5 to 35.6]
Statistical Analysis 5: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Checklist use; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 413, 95% CI 2-sided [65.8 to 2589]

17. Other Pre Specified Outcome: Count of Participants Where Essential Birth Practices Were Observed Just Before Pushing, 2 Months Post-intervention Start
Description: Birth attendant's rate of completion of "Process measures" resulting from Safe Childbirth Checklist program will be assessed in a sample of total birth events at 2 months after the intervention is introduced to intervention facilities. The below measures reflect the essential birth practices performed at the time of labor just before pushing, 2 months post-intervention start.
Time Frame: 2 months post-intervention start
Population: The denominator for this analysis is all women who were observed at the time of labor just before pushing, 2 months post-intervention start in the site.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 1039 | 1130
Participants
  Hand hygiene | 367 | 7
  No oxytocin given before delivery | 704 | 333
  Clean towel available | 874 | 166
  Clean scissors or blade available | 843 | 847
  Cord tie available | 1035 | 1122
  Mucus extractor available | 990 | 1057
  Neonatal bag and mask available | 991 | 1109
  Pads available | 965 | 502
  Checklist Use | 255 | 1
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Hand hygiene; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 53.3, 95% CI 2-sided [13.1 to 217]
Statistical Analysis 2: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; No oxytocin given before delivery; Test type: Superiority; p = 0.007, Chi-squared, Corrected; Risk Ratio (RR) = 2.3, 95% CI 2-sided [1.3 to 4.2]
Statistical Analysis 3: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Clean towel available; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 5.7, 95% CI 2-sided [2.7 to 12.1]
Statistical Analysis 4: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Clean scissors or blade available; Test type: Superiority; p = 0.72, Chi-squared, Corrected; Risk Ratio (RR) = 1.1, 95% CI 2-sided [0.7 to 1.7]
Statistical Analysis 5: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Cord tie available; Test type: Superiority; p = 0.48, Chi-squared, Corrected; Risk Ratio (RR) = 1.0, 95% CI 2-sided [1.0 to 1.0]
Statistical Analysis 6: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Mucus extractor available; Test type: Superiority; p = 0.73, Chi-squared, Corrected; Risk Ratio (RR) = 1.0, 95% CI 2-sided [0.9 to 1.1]
Statistical Analysis 7: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Neonatal bag and mask available; Test type: Superiority; p = 0.56, Chi-squared, Corrected; Risk Ratio (RR) = 1.0, 95% CI 2-sided [0.9 to 1.1]
Statistical Analysis 8: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Pads available; Test type: Superiority; p = 0.005, Chi-squared, Corrected; Risk Ratio (RR) = 2.1, 95% CI 2-sided [1.3 to 3.5]
Statistical Analysis 9: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Checklist use; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 185, 95% CI 2-sided [19.7 to 1738]

18. Other Pre Specified Outcome: Count of Participants Where Essential Birth Practices Were Observed Within One Minute After Delivery, 2 Months Post-intervention Start
Description: Birth attendant's rate of completion of "Process measures" resulting from Safe Childbirth Checklist program will be assessed in a sample of total birth events at 2 months after the intervention is introduced to intervention facilities. The below measures reflect the essential birth practices performed at the time within one minute after the woman's delivery, 2 months post-intervention start.
Time Frame: 2 months post-intervention start
Population: The denominator for this analysis is all women who were observed within one minute after delivery, 2 months post-intervention start in the site.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 1038 | 1129
Participants
  Oxytocin Administered | 825 | 231
  Neonatal bag used | 47 | 82
  Birth companion present | 1037 | 1125
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Oxytocin administered; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 3.9, 95% CI 2-sided [2.1 to 7.2]
Statistical Analysis 2: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Neonatal bag used; Test type: Superiority; p = 0.25, Chi-squared, Corrected; Risk Ratio (RR) = 0.6, 95% CI 2-sided [0.3 to 1.4]
Statistical Analysis 3: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Birth attendant present; Test type: Superiority; p = 0.25, Chi-squared, Corrected; Risk Ratio (RR) = 1.0, 95% CI 2-sided [1.0 to 1.0]

19. Other Pre Specified Outcome: Count of Participants Where Essential Birth Practices Were Observed Within One Hour After Delivery, 2 Months Post-intervention Start
Description: Birth attendant's rate of completion of "Process measures" resulting from Safe Childbirth Checklist program will be assessed in a sample of total birth events at 2 months after the intervention is introduced to intervention facilities. The below measures reflect the essential birth practices performed within one hour after delivery, 2 months post-intervention start.
Time Frame: 2 months post-intervention start
Population: The denominator for this analysis is all women who were observed at one hour after delivery, 2 months post-intervention start in the site.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 1006 | 1102
Participants
  Newborn weight taken | 906 | 884
  Newborn temperature taken | 433 | 1
  Skin-to-skin care initiated at birth | 794 | 119
  Skin-to-skin care maintained for 1 hr | 194 | 5
  Initiation of breast-feeding | 700 | 39
  Checklist use | 747 | 0
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Newborn weight taken; Test type: Superiority; p = 0.25, Chi-squared, Corrected; Risk Ratio (RR) = 1.1, 95% CI 2-sided [0.9 to 1.4]
Statistical Analysis 2: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Newborn temperature taken; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 317, 95% CI 2-sided [50.4 to 1989]
Statistical Analysis 3: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Skin-to-skin care initiated at birth; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 7.3, 95% CI 2-sided [2.4 to 22.0]
Statistical Analysis 4: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Skin-to-skin care maintained for 1 hr; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 38.7, 95% CI 2-sided [7.7 to 194]
Statistical Analysis 5: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Initiation of breast-feeding; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 19.4, 95% CI 2-sided [11.4 to 33.2]
Statistical Analysis 6: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Checklist use; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Other = 0 — The relative risk could not be calculated owing to 100% or 0% values in one group

20. Other Pre Specified Outcome: Count of Participants Where Essential Birth Practices Were Observed at Anytime During Delivery, 2 Months Post-intervention Start
Description: Birth attendant's rate of completion of "Process measures" resulting from Safe Childbirth Checklist program will be assessed in a sample of total birth events at 2 months after the intervention is introduced to intervention facilities. The below measures reflect the essential birth practices performed at anytime during the observation period of the woman's delivery, 2 months post-intervention start.
Time Frame: 2 months post-intervention start
Population: The denominator for this analysis is all women who were observed at any time during delivery, 2 months post-intervention start in the site.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 1259 | 1304
Participants
  Maternal temperature taken | 792 | 4
  Maternal blood pressure taken | 854 | 89
  Mother given magnesium sulfate | 1 | 3
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Maternal temperature taken; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 182, 95% CI 2-sided [33.5 to 993]
Statistical Analysis 2: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Maternal blood pressure taken; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 9.9, 95% CI 2-sided [3.8 to 25.8]
Statistical Analysis 3: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Mother given magnesium sulfate; Test type: Superiority; p = 0.30, Chi-squared, Corrected; Risk Ratio (RR) = 0.4, 95% CI 2-sided [0.1 to 2.1]

21. Other Pre Specified Outcome: Mean Number of 18 Essential Birth Practices Performed at 12 Months Post-intervention Start
Description: Birth attendant's rate of completion of "Process measures" resulting from Safe Childbirth Checklist program will be assessed in a sample of total birth events at 12 months after the intervention is introduced to intervention facilities. The below measures reflect the mean number of 18 essential birth practices performed across the intervention versus control facilities at 12 months post-intervention start.
Time Frame: 12 months post-intervention start
Population: The denominator for this analysis is all women who were observed for at least one pause point 12 months post-intervention start in the site.
Measure: Mean (95% Confidence Interval); unit: essential birth practices performed
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 1127 | 1198
essential birth practices performed | 11.1 [10.4 to 11.8] | 7.9 [7.4 to 8.4]
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Other = 0

22. Other Pre Specified Outcome: Count of Participants Where Essential Birth Practices Were Observed at Admission, 12 Months Post-intervention Start
Description: Birth attendant's rate of completion of "Process measures" resulting from Safe Childbirth Checklist program will be assessed in a sample of total birth events at 12 months after the intervention is introduced to intervention facilities. The below measures reflect the essential birth practices performed at the time of the woman's admission to the facility, 12 months post-intervention start.
Time Frame: 12 months post-intervention start
Population: The denominator for this analysis is all women who were observed at admission, 12 months post-intervention start in the site.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 1007 | 1009
Participants
  Birth companion present | 1004 | 1006
  Maternal blood pressure taken | 219 | 11
  Maternal temperature taken | 153 | 0
  Partography started | 7 | 0
  Checklist use | 175 | 0
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Birth companion present; Test type: Superiority; p = 1.00, Chi-squared, Corrected; Risk Ratio (RR) = 1.0, 95% CI 2-sided [1.0 to 1.0]
Statistical Analysis 2: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Maternal blood pressure taken; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 19.1, 95% CI 2-sided [7.9 to 46.5]
Statistical Analysis 3: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Maternal temperature taken; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Other = 0 — The relative risk could not be calculated due to 100% or 0% values in one group
Statistical Analysis 4: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Partography started; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Other = 0 — The relative risk could not be calculated owing to 100% or 0% values in one group
Statistical Analysis 5: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Checklist use; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Other = 0 — The relative risk could not be calculated owing to 100% or 0% values in one group

23. Other Pre Specified Outcome: Count of Participants Where Essential Birth Practices Were Observed Just Before Pushing, 12 Months Post-intervention Start
Description: Birth attendant's rate of completion of "Process measures" resulting from Safe Childbirth Checklist program will be assessed in a sample of total birth events at 12 months after the intervention is introduced to intervention facilities. The below measures reflect the essential birth practices performed at the time just before pushing, 12 months post-intervention start
Time Frame: 12 months post-intervention start
Population: The denominator for this analysis is all women who were observed at the time just before pushing, 12 months post-intervention start in the site.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 1018 | 1042
Participants
  Hand hygiene | 126 | 6
  No oxytocin given before delivery | 527 | 263
  Clean towel available | 721 | 314
  Clean scissors or blade available | 1004 | 1008
  Cord tie available | 1009 | 1039
  Mucus extractor available | 999 | 1000
  Neonatal bag and mask available | 1017 | 1036
  Pads available | 768 | 559
  Checklist Use | 55 | 1
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Hand hygiene; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 19.9, 95% CI 2-sided [6.6 to 60.4]
Statistical Analysis 2: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; No oxytocin given before delivery; Test type: Superiority; p = 0.04, Chi-squared, Corrected; Risk Ratio (RR) = 2.1, 95% CI 2-sided [1.0 to 4.1]
Statistical Analysis 3: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Clean towel available; Test type: Superiority; p = 0.006, Chi-squared, Corrected; Risk Ratio (RR) = 2.4, 95% CI 2-sided [1.3 to 4.3]
Statistical Analysis 4: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Clean scissors or blade available; Test type: Superiority; p = 0.34, Chi-squared, Corrected; Risk Ratio (RR) = 1.0, 95% CI 2-sided [1.0 to 1.1]
Statistical Analysis 5: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Cord tie available; Test type: Superiority; p = 0.25, Chi-squared, Corrected; Risk Ratio (RR) = 1.0, 95% CI 2-sided [1.0 to 1.0]
Statistical Analysis 6: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Mucus extractor available; Test type: Superiority; p = 0.50, Chi-squared, Corrected; Risk Ratio (RR) = 1.0, 95% CI 2-sided [1.0 to 1.1]
Statistical Analysis 7: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Neonatal bag and mask available; Test type: Superiority; p = 0.32, Chi-squared, Corrected; Risk Ratio (RR) = 1.0, 95% CI 2-sided [1.0 to 1.0]
Statistical Analysis 8: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Pads available; Test type: Superiority; p = 0.11, Chi-squared, Corrected; Risk Ratio (RR) = 1.4, 95% CI 2-sided [0.9 to 2.1]
Statistical Analysis 9: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Checklist available; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 37.9, 95% CI 2-sided [7.3 to 196]

24. Other Pre Specified Outcome: Count of Participants Where Essential Birth Practices Were Observed Within One Minute After Delivery, 12 Months Post-intervention Start
Description: Birth attendant's rate of completion of "Process measures" resulting from Safe Childbirth Checklist program will be assessed in a sample of total birth events at 12 months after the intervention is introduced to intervention facilities. The below measures reflect the essential birth practices performed within one minute after delivery, 12 months post-intervention start
Time Frame: 12 months post-intervention start
Population: The denominator for this analysis is all women who were observed within one minute after delivery, 12 months post-intervention start in the site.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 1019 | 1041
Participants
  Oxytocin Administered | 549 | 154
  Neonatal bag used | 30 | 49
  Birth companion present | 1016 | 1035
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Oxytocin administered; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 3.6, 95% CI 2-sided [1.8 to 7.5]
Statistical Analysis 2: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Neonatal bag used; Test type: Superiority; p = 0.19, Chi-squared, Corrected; Risk Ratio (RR) = 0.6, 95% CI 2-sided [0.3 to 1.3]
Statistical Analysis 3: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Birth companion present; Test type: Superiority; p = 0.50, Chi-squared, Corrected; Risk Ratio (RR) = 1.0, 95% CI 2-sided [1.0 to 1.0]

25. Other Pre Specified Outcome: Count of Participants Where Essential Birth Practices Were Observed Within One Hour After Delivery, 12 Months Post-intervention Start
Description: Birth attendant's rate of completion of "Process measures" resulting from Safe Childbirth Checklist program will be assessed in a sample of total birth events at 12 months after the intervention is introduced to intervention facilities. The below measures reflect the essential birth practices performed within one hour after delivery, 12 months post-intervention start
Time Frame: 12 months post-intervention start
Population: The denominator for this analysis is all women who were observed within one hour after delivery, 12 months post-intervention start in the site.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 1000 | 1014
Participants
  Newborn weight taken | 947 | 843
  Newborn temperature taken | 225 | 2
  Skin-to-skin care initiated at birth | 685 | 84
  Skin-to-skin care maintained for 1 hr | 51 | 0
  Initiation of breast-feeding | 369 | 47
  Checklist use | 351 | 0
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Newborn weight taken; Test type: Superiority; p = 0.08, Chi-squared, Corrected; Risk Ratio (RR) = 1.1, 95% CI 2-sided [1.0 to 1.3]
Statistical Analysis 2: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Newborn temperature taken; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 91.5, 95% CI 2-sided [11.0 to 758]
Statistical Analysis 3: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Skin-to-skin care initiated at birth; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 8.2, 95% CI 2-sided [2.5 to 27.5]
Statistical Analysis 4: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Skin-to-skin care maintained for 1 hr; Test type: Superiority; p = 0.01, Chi-squared, Corrected; Other = 0 — The relative risk could not be calculated owing to 100% or 0% values in one group
Statistical Analysis 5: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Initiation of breast-feeding; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 7.9, 95% CI 2-sided [3.7 to 16.7]
Statistical Analysis 6: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Checklist use; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Other = 0 — The relative risk could not be calculated owing to 100% or 0% values in one group

26. Other Pre Specified Outcome: Count of Participants Where Essential Birth Practices Were Observed at Anytime, 12 Months Post-intervention Start
Description: Birth attendant's rate of completion of "Process measures" resulting from Safe Childbirth Checklist program will be assessed in a sample of total birth events at 12 months after the intervention is introduced to intervention facilities. The below measures reflect the essential birth practices performed at any time during the observation period, 12 months post-intervention start.
Time Frame: 12 months post-intervention start
Population: The denominator for this analysis is all women who were observed at anytime, 12 months post-intervention start in the site.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Health Facility Participants: Women at intervention facilities who registered for labor and delivery, eligible for inclusion, and who provided consent for observation.
  Intervention Health Facilities received the WHO Safe Childbirth Checklist Program.
  WHO Safe Childbirth Checklist Program: The IHF group will receive the WHO Safe Childbirth Checklist Program designed to maximize likelihood of effective and sustained uptake of the program by birth attendants in the designated facilities. The program includes three key implementation steps that involve: engagement of leadership and clinicians at the state, district, and local levels, a formal launch to introduce the Checklist, and support through peer coaching and data feedback. The intervention facilities will also receive a standardized maternity register to ensure appropriate data collection.
- Control Health Facility Participants: Women at control health facilities who registered for labor and delivery, eligible for inclusion, and who provided consent for observation.
  Matched control facilities provided comparison for intervention facilities.
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
Number analyzed (Participants) | 1127 | 1198
Participants
  Maternal temperature taken | 343 | 0
  Maternal blood pressure taken | 425 | 35
  Mother given magnesium sulfate | 1 | 1
Statistical Analysis 1: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Maternal temperature taken; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Other = 0 — The relative risk could not be calculated owing to 100% or 0% values in one group
Statistical Analysis 2: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Maternal blood pressure taken; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Risk Ratio (RR) = 12.7, 95% CI 2-sided [4.7 to 34.3]
Statistical Analysis 3: Comparison: Intervention Health Facility Participants vs Control Health Facility Participants; Mother given magnesium sulfate; Test type: Superiority; p = 0.95, Chi-squared, Corrected; Risk Ratio (RR) = 1.1, 95% CI 2-sided [0.2 to 6.6]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for occurrence and reporting throughout the duration of the study period (2 years).
Description: Maternal & neonatal mortality were measured as outcomes, not as adverse events. No adverse events such as death or morbidity were linked to direct effect of the trial. Our adverse events included loss of a consent form or a breach of PHI.
  While our outcomes denominators reflect either the woman/newborn dyad or women only, this denominator includes all individual mothers plus all individual newborns enrolled in the trial, in order to obtain an all cause mortality count.
Arm/Group | Intervention Health Facility Participants | Control Health Facility Participants
All-Cause Mortality (participants affected / at risk) | 3917/159587 | 3677/154684
Serious Adverse Events (participants affected / at risk) | 0/159587 | 0/154684
Other Adverse Events (participants affected / at risk) | 0/159587 | 0/154684

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/52/NCT02148952/Prot_SAP_000.pdf